CLINICAL TRIAL: NCT04078373
Title: Assessment and Treatment of Urinary Disorders in Patients in the Subacute Phase After Stroke
Brief Title: Urinary Disorders in Subacute Patients After Stroke
Acronym: UIMK
Status: Recruiting | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Other Study IDs: URIS201901
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Urinary Incontinence
Keywords: stroke; inpatient rehabilitation; urinary disorders; treatment
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Urinary Incontinence; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without urinary disorders: Subacute stroke patients without urinary disorders
- With urinary disorders: Subacute stroke patients with urinary disorders
  Interventions: Behavioral: Immediate urination; Behavioral: Bladder diary

INTERVENTIONS:
Behavioral: Immediate urination — Patients with decreased cognitive ability will be taught to immediately go to the toilet upon feeling the urge to urinate and to be independent in urinating.
  Groups: With urinary disorders
Behavioral: Bladder diary — Patients with normal cognitive abilities will be instructed to go to the toilet every 2-3 hours regardless of the urge to urinate
  Groups: With urinary disorders

SUMMARY:
This observational study will address urinary disorders in subacute stroke patients. Patients without and with urinary disorders will be compared, and treatment outcome will be assessed among the latter.

DETAILED DESCRIPTION:
This prospective observational study will include 100 patients after first ischaemic or hemorrhagic stroke directly transferred from an acute hospital to our Institute for inpatient rehabilitation. Within admission assessment, patients will be classified according to stroke type, stroke localisation and time since stroke. Comorbidities will be recorded and associated neurological deficits will be assessed. Post mictional residue will be determined in all patients one day after admission. The patients with urinary disorders will be treated according to the published official protocol, either using the immediate urination approach or the bladder diary approach. Continence will be regularly assessed by the nursing staff. Urination-disorder-related complications (pressure ulcers, falls and urinary infections), drug therapy and the use of continence aids will also be followed.

ELIGIBILITY:
Inclusion Criteria:

* subacute patients after ischaemic or hemorrhagic stroke;
* direct transfer from acute hospital to complex inpatient rehabilitation at our Institute.

Exclusion Criteria:

* incontinence before stroke;
* previous brain injury or other brain disease;
* previous bladder or prostate surgery;
* inability to ambulate before stroke;
* terminal disease with expected survival less than three months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subacute patients after ischaemic or hemorrhagic stroke directly transferred from an acute hospital to complex inpatient rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Degree of urinary continence | Through study completion, for an average of 6 weeks
  Urinary continence will be assessed daily by the nursing staff as either complete, partial or incontinence

SECONDARY OUTCOMES:
Presence of urinary-disorders-related complications | Through study completion, for an average of 6 weeks
  Pressure ulcers, falls and urinary infections caused by urinary disorders will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nataša Bizovičar, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No